CLINICAL TRIAL: NCT04027777
Title: Single-center Prospective Observational Study to Validate the Performance of the Aktiia Optical Blood Pressure Monitoring (OBPM) Device at the Wrist Against Double Auscultation
Brief Title: Aktiia OPBM Single-center Prospective Observational Study Against Double Auscultation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aktiia SA (Industry)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: OBPM_Ambulatory2019
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aktiia.product-P0 (Experimental): Main study arm including 85 subjects
  Interventions: Device: Aktiia.product-P0
- Aktiia.product-P0 Diabetics (Experimental): Second study arm including 40 diabetic patients
  Interventions: Device: Aktiia.product-P0
- Aktiia.product-P0 Aged (Experimental): Thirs study arm including 40 patients aged 65+
  Interventions: Device: Aktiia.product-P0

INTERVENTIONS:
Device: Aktiia.product-P0 — The optical signals at the wrist are recorded non-invasively by means of the Aktiia.product-P0 investigational device. The BP measurements are further determined from these optical signals and are compared to the reference double auscultation BP readings. A reference-control volume clamp BP reading is recorded simultaneously.

SUMMARY:
Single-centre prospective observational study to validate the performance of the Aktiia SA optical blood pressure monitoring (OBPM) device at the wrist against blood pressure measurements obtained by double auscultation at the upper arm during four weeks

DETAILED DESCRIPTION:
According to the World Health Organization, by 2025 hypertension will affect 1.5 billion adults worldwide. Half of the adult population is not diagnosed, and half of the treated population is not at the defined target of BP. Widespread use of out of office BP measurement is one of the proposed strategies to fight against hypertension worldwide.

The current Ambulatory Blood Pressure Monitoring or Home Blood Pressure Monitoring are performed with a cuff placed around the arm. This 110-year-old technology is not only uncomfortable for the patient but can also result in a number of overestimated readings due to the stress induced while inflating the cuff.

Aktiia S.A. has developed an intermittent automated non-invasive cuffless blood pressure monitor determining over a series of cardiac cycles the values of the systolic blood pressure, the diastolic blood pressure and the heart rate. This miniature device is comfortably positioned with a bracelet on a user's wrist. The optical sensors integrated within the device exploit the principle of reflection photoplethysmography (PPG) to capture the user's skin pulsatility (change of arterial diameter occurring at each heartbeat). Aktiia OBPM algorithms are further applied to the recorded PPG signal to determine user's blood pressure and heart rate.

Because the measurement relies on optical sensors, and not on pneumatic cuffs, Aktiia OBPM device provides an increased overall comfort to the patient throughout the monitoring, does not induce sleep arousal during the night measurements and decreases the false positive readings induced by the stress associated with the cuff inflation. Aktiia OBPM device is intended to be used in the long term, as compared to one-day or one-week use of Ambulatory Blood Pressure Monitors.

This study over several visits has been designed to assess both the accuracy and the stability of the Aktiia OBPM. The automaticity of the measurement when performed in different body positions and upon aerobic exercise was also evaluated.

By demonstrating both the accuracy and the stability of the measurements that can be performed in different body positions with a comfortable and miniature Aktiia OBPM device, Aktiia SA aims to make one step further in facilitating blood pressure measurement and monitoring in the out-of-clinic scenarios and integrating blood pressure monitoring into user's daily life. The diagnosis and treatment of hypertension in ambulatory settings is expected to largely benefit from these advancements

ELIGIBILITY:
ARM1

Inclusion Criteria:

* Adult subjects (aged between 21 and 65 years old)
* Subjects fluent in written and spoken French
* Subjects agreeing to attend the totality of 4 visits
* Subjects that have signed the informed consent form

Exclusion Criteria:

* Subjects with tachycardia (heart rate at rest > 120bpm)
* Subjects with atrial fibrillation
* Subjects with diabetes
* Subjects with renal dysfunctions (eGFR < 60mL/min/1.73 m2)
* Subjects with hyper-/hypothyroidism
* Subjects with pheochromocytoma
* Subjects with Raynaud's disease
* Subjects with trembling and shivering
* Subjects with interarm systolic difference > 15 mmHg
* Subjects with interarm diastolic difference > 10 mmHg
* Subjects with arm paralysis
* Women in known pregnancy
* Subjects with an arteriovenous fistula
* Subjects with arm amputations
* Subjects with the upper arm circumference > 64 cm
* Subjects with the wrist circumference > 22 cm (limitation due Aktiia.bracelet-P0 size)
* Subjects with the central phalanx of the middle finger circumference > 71 mm or < 43 mm
* Subjects with the exfoliative skin diseases (limitation due to participant discomfort)
* Subjects with lymphoedema (limitation due to participant discomfort)

ARM2

Inclusion Criteria:

* Adult subjects (aged between 21 and 65 years old)
* Subjects fluent in written and spoken French
* Subjects agreeing to attend the totality of 4 visits
* Subjects that have signed the informed consent form

Exclusion Criteria:

* Subjects with tachycardia (heart rate at rest > 120bpm)
* Subjects with atrial fibrillation
* Subjects with hyper-/hypothyroidism
* Subjects with pheochromocytoma
* Subjects with Raynaud's disease
* Subjects with trembling and shivering
* Subjects with interarm systolic difference > 15 mmHg
* Subjects with interarm diastolic difference > 10 mmHg
* Subjects with arm paralysis
* Women in known pregnancy
* Subjects with an arteriovenous fistula
* Subjects with arm amputations
* Subjects with the upper arm circumference > 64 cm
* Subjects with the wrist circumference > 22 cm (limitation due Aktiia.bracelet-P0 size)
* Subjects with the central phalanx of the middle finger circumference > 71 mm or < 43 mm
* Subjects with the exfoliative skin diseases (limitation due to participant discomfort)
* Subjects with lymphoedema (limitation due to participant discomfort)

ARM3

Inclusion Criteria:

* Adult subjects (aged between 65 and 85 years old)
* Subjects fluent in written and spoken French
* Subjects agreeing to attend the totality of 4 visits
* Subjects that have signed the informed consent form

Exclusion Criteria:

* Subjects with tachycardia (heart rate at rest > 120bpm)
* Subjects with atrial fibrillation
* Subjects with diabetes
* Subjects with renal dysfunctions (eGFR < 60mL/min/1.73 m2)
* Subjects with hyper-/hypothyroidism
* Subjects with pheochromocytoma
* Subjects with Raynaud's disease
* Subjects with trembling and shivering
* Subjects with interarm systolic difference > 15 mmHg
* Subjects with interarm diastolic difference > 10 mmHg
* Subjects with arm paralysis
* Women in known pregnancy
* Subjects with an arteriovenous fistula
* Subjects with arm amputations
* Subjects with the upper arm circumference > 64 cm
* Subjects with the wrist circumference > 22 cm (limitation due Aktiia.bracelet-P0 size)
* Subjects with the central phalanx of the middle finger circumference > 71 mm or < 43 mm
* Subjects with the exfoliative skin diseases (limitation due to participant discomfort)
* Subjects with lymphoedema (limitation due to participant discomfort)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure absolute Mean Error | Up to four weeks
  The absolute value of the mean of the differences between Reference and Aktiia.product-P0 blood pressure determinations
Blood Pressure standard Deviation of the Error | Up to four weeks
  The standard deviation of the differences between Reference and Aktiia.product-P0 determinations

SECONDARY OUTCOMES:
Heart Rate root-mean-square error | Up to four weeks
  The root-mean-square difference between the Aktiia.product-P0 heart rate determinations and the Reference method

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire Wuerzner, MD, Principal Investigator — CHUV
Locations (1):
- University of Lausanne Hospitals, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Theiler K, Sola J, Damianaki A, Pfister A, Almeida TP, Alexandre J, Vermare P, Wuerzner G. Performance of the Aktiia optical blood pressure measurement device in the elderly: a comparison with double blinded auscultation in different body positions. Blood Press. 2023 Dec;32(1):2281320. doi: 10.1080/08037051.2023.2281320. Epub 2023 Nov 16. PMID 37971487
- See also: Sponsor website — http://www.aktiia.com